CLINICAL TRIAL: NCT02441244
Title: Probiotic Visbiome for Inflammation and Translocation in HIV I (PROOV IT I)
Brief Title: Probiotic Visbiome for Inflammation and Translocation in HIV Ι
Acronym: PROOV IT I
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment potential impaired by shift in clinical care whereby practically all HIV patients receive standard treatment as soon as possible after HIV diagnosis
Sponsor: University Health Network, Toronto (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTNPT 022A
Record Dates: First submitted 2015-04-23; First posted 2015-05-12 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic Group (Experimental): Visbiome experimental group (900 billion bacteria daily; 2 sachets daily)
  Interventions: Drug: Visbiome
- Placebo Group (Placebo Comparator): Placebo comparator group
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Visbiome — Visbiome probiotic
  Arms: Probiotic Group
Other: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
Modern antiretroviral therapy (ART) has transformed the clinical care and lived experience of HIV infection. However, increased rates of adverse health conditions that are related to immune activation, such as cardiovascular disease (CVD) and neurodegenerative disease in ART-treated individuals persist. An important cause of this inflammation is the gut CD4 T cell loss and the "leaking" or translocation of luminal gut bacteria and other microbes across the bowel wall and into the bloodstream.

The use of complementary and alternative therapies is common among people living with HIV, however their efficacy has generally not been well demonstrated. Probiotics are live microbes that may provide a health benefit to the host and the investigators believe that the simultaneous use of probiotics along with antiretroviral therapy (ART) will improve gut CD4 T cell restoration and function and therefore reduce microbial translocation and immune activation.

Probiotic Visbiome consists of a high potency blend of eight different probiotics. The precise mechanism of action of Visbiome is unknown, but preclinical studies have shown that Visbiome may modulate the immune response towards a phenotype that is associated with reduce inflammation, and Visbiome was also protective in a non-human primate model of SIV infection. Therefore, we believe that the "beneficial" bacteria from Visbiome will accelerate the normalization of gut immune cells and function in HIV-infected individuals as they start ART. Early resolution of gut immune cells may normalize microbial translocation and immune activation and will reduce the rates of HIV-associated comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Male adult (age >18 years)
* Antiretroviral therapy-naïve
* Ability to provide informed consent
* HIV-1 viral load ≥1,000 copies/ml

Exclusion Criteria:

* Current alcohol or substance use judged by the Investigator to potentially interfere with participant study compliance
* Taking pharmaceutical grade probiotics
* Any of the following abnormal laboratory results in screening:

  * Hemoglobin <85 g/L
  * Neutrophil count <750 cells/μl
  * Platelet count <50,000 cells/μl
  * AST or ALT >5X the upper limit of normal
* Malignancy
* Colitis
* Liver fibrosis (decompensated cirrhosis), portal hypertension or clinical hepatitis
* Other significant underlying disease (non-HIV-1) that might impinge upon disease progression or death

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-11-15 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
Blood immune activation | 24 weeks
  Percent of blood immune activation (coexpression of CD38 and HLA-DR) on CD8 T cells at week 24 in participants randomized to probiotic Visbiome versus the placebo arm

SECONDARY OUTCOMES:
Level of microbial translocation (including LPS and sCD14) | 24 weeks
Plasma level of inflammation and coagulation (including IL-6, D-dimer and CRP) | 24 weeks
Number and function of gut immune cells (including CD4 T cell subsets) | 24 weeks
Intestinal permeability (Lac/Mac ratio) | 24 weeks
Microbiome analysis by 16s rRNA bacterial DNA isolated from gut tissue and anal swabs | 24 weeks
Gut HIV DNA levels | 24 weeks
Canadian Diet History Questionnaire | 24 weeks
Safety assessed by AE monitoring and participant questionnaire | 24 weeks
Tolerability of Visbiome assessed by AE monitoring and participant questionnaire | 24 weeks
Adherence to probiotic Visbiome assessed by participant questionnaire and sachet count | 24 weeks

OTHER OUTCOMES:
Metabolomic measurements: vitamin D levels, glucose measurements, insulin levels and lipid profiling | 24 weeks
Bacterial community diversity, determined by 16s rRNA gene sequencing of penile swabs | 24 weeks
Bacterial community composition, determined by 16s rRNA gene sequencing of penile swabs | 24 weeks
Blood immune activation (open-label) | 48 weeks
  Percent of blood immune activation (coexpression of CD38 and HLA-DR) on CD8 T cells at week 24 in participants randomized to probiotic Visbiome versus the placebo arm
Level of microbial translocation (including LPS and sCD14) (open-label) | 48 weeks
Plasma levels of inflammation and coagulation (including IL-6, D-dimer and CRP) (open-label) | 48 weeks
Number and function of gut immune cells (including CD4 T cell subsets) (open-label) | 48 weeks
Intestinal permeability (Lac/Man) (open-label) | 48 weeks
Microbiome analysis by 16s rRNA bacterial DNA isolated from penile swabs (open-label) | 48 weeks
Gut HIV DNA levels (open-label) | 48 weeks
Canadian Diet History Questionnaire (open-label) | 48 weeks
Safety (open-label) assessed by AE monitoring and participant questionnaire | 48 weeks
Tolerability of Visbiome (open-label) assessed by AE monitoring and participant questionnaire | 48 weeks
Adherence to probiotic Visbiome (open-label) assessed by participant questionnaire and sachet count | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Kaul, MD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Maple Leaf Medical Clinic, Toronto, Ontario
  - Toronto General Hospital, UHN, Toronto, Ontario